CLINICAL TRIAL: NCT00000545
Title: PATHWAYS--FULL SCALE STUDY
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Purpose: Prevention
Other Study IDs: 88; U01HL050869 (NIH); U01HL050907 (NIH); U01HL050905 (NIH); U01HL050885 (NIH)
Record Dates: First submitted 1999-10-27; First posted 1999-10-28 (Estimated); Last update posted 2016-07-29 (Estimated); Status verified 2005-12

CONDITIONS: Cardiovascular Diseases; Sedentary Behaviors; Obesity
MeSH Terms: conditions — Cardiovascular Diseases; Sedentary Behavior; Obesity | interventions — Exercise; Diet

INTERVENTIONS:
Behavioral: exercise
Behavioral: diet

SUMMARY:
To implement a culturally appropriate school-based, multicenter, randomized trial that promotes healthful eating behaviors and increases physical activity to prevent obesity in pre-adolescent upper elementary American Indian students.

DETAILED DESCRIPTION:
BACKGROUND:

The American Indian population, including American Indians and Alaska Natives, totals nearly 1.5 million from over 500 tribes and nearly 300 reservations and Alaska Native villages. Earlier in this century, heart disease was rarely noted in American Indians, but in the past decade, cardiovascular disease has become the leading cause of death in American Indians. Several factors may be responsible for this increase: a decreasing incidence of infectious disease, an increasing incidence of diabetes mellitus, and an increasing incidence of obesity. Previous research on non-Indian populations indicates that obesity is an independent risk factor for cardiovascular disease and that it is associated with increases in other cardiovascular disease risk factors such as high blood pressure, diabetes, and low high density lipoprotein cholesterol levels. The high prevalence of obesity among American Indians, coupled with its role as a risk factor for hypertension, coronary heart disease, and diabetes, suggests that a reduction in the average weight of young American Indians would improve their health. Reduction of the prevalence of obesity in American Indians has been designated as a goal for improving the health of this minority population and reducing health disparities in our nation.

The successful 4-1/2 year feasibility study was followed by the full-scale randomized trial involving 1,700 American Indian elementary schoolchildren. Schools were the unit of randomization.

The initiative was developed as a result of consultations with the NHLBI Ad Hoc Committee on Minority Populations, the Conference on Obesity and Cardiovascular Disease in Minority Populations, and the Indian Health Service. The need for the study was reinforced by the preliminary data from the Strong Heart Study confirming the high prevalence of obesity in American Indians. The initiative was approved by the Clinical Applications and Prevention Advisory Committee in February 1992 and given concept clearance by the National Heart, Lung, and Blood Advisory Council in May 1992.

DESIGN NARRATIVE:

The Feasibility Phase of the trial was completed in 1995. The organizational structure has been established, validation studies to determine an endpoint and formative assessment of the tribe communities was completed. Intervention including classroom curriculum, food service, physical activity family component and for the measurement methods including obesity, physical activity, diet intake, knowledge, attitudes and behavior, and process evaluation were completed.

The full-scale trial started in September 1996. The primary aim was to test the effectivenes of a culturally appropriate school-based intervention that promoted increased physical activity and healthful eating behaviors to prevent obesity in American Indian upper elementary school children. The primary outcome was percent body fat after three years of intervention. The major hypothesis was that intervention would result in an absolute difference of 3 percent body fat between the control and intervention schools. All students enrolled in the second grade in the participating schools during Spring, 1997 participated in the baseline survey. Baseline measurements were performed at the end of second grade so that the intervention could begin at the start of third grade. The intervention lasted for three years. A single cohort of children progressed through third, fourth, and fifth grades. Schools were the unit of randomization. Forty-one schools in four centers were stratified within each field center on median percent body fat (PBF) at the end of second grade using data from the baseline measurement. Schools within a field center were then ranked on median PBF. Once stratified, the coordinating center randomly assigned half the schools within each stratum to intervention (21) and half to control (20).

The study completion date listed in this record was obtained from the "End Date" entered in the Protocol Registration and Results System (PRS) record.

ELIGIBILITY:
Cohort of pre-adolescent American Indian boys and girls followed in grades 3-5.

Ages: 7 Years to 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Dates: Start 1993-09; Study Completion 2002-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: H. Stevens — University of North Carolina

REFERENCES:
- [Background] Prevention of obesity in American Indian children: the Pathways study. Am J Clin Nutr. 1999 Apr;69(4 Suppl):745S-824S. doi: 10.1093/ajcn/69.4.745S. No abstract available. PMID 10195596
- [Background] Caballero B: Introduction. Am J Clin Nutr, 69: 745S-746S, 1999.
- [Background] Story M, Evans M, Fabsitz RR, Clay TE, Holy Rock B, Broussard B. The epidemic of obesity in American Indian communities and the need for childhood obesity-prevention programs. Am J Clin Nutr. 1999 Apr;69(4 Suppl):747S-754S. doi: 10.1093/ajcn/69.4.747S. PMID 10195597
- [Background] Davis CE, Hunsberger S, Murray DM, Fabsitz RR, Himes JH, Stephenson LK, Caballero B, Skipper B. Design and statistical analysis for the Pathways study. Am J Clin Nutr. 1999 Apr;69(4 Suppl):760S-763S. doi: 10.1093/ajcn/69.4.760S. PMID 10195599
- [Background] Lohman TG, Caballero B, Himes JH, Hunsberger S, Reid R, Stewart D, Skipper B. Body composition assessment in American Indian children. Am J Clin Nutr. 1999 Apr;69(4 Suppl):764S-766S. doi: 10.1093/ajcn/69.4.764S. PMID 10195600
- [Background] Gittelsohn J, Evans M, Story M, Davis SM, Metcalfe L, Helitzer DL, Clay TE. Multisite formative assessment for the Pathways study to prevent obesity in American Indian schoolchildren. Am J Clin Nutr. 1999 Apr;69(4 Suppl):767S-772S. doi: 10.1093/ajcn/69.4.767S. PMID 10195601
- [Background] Stevens J, Cornell CE, Story M, French SA, Levin S, Becenti A, Gittelsohn J, Going SB, Reid R. Development of a questionnaire to assess knowledge, attitudes, and behaviors in American Indian children. Am J Clin Nutr. 1999 Apr;69(4 Suppl):773S-781S. doi: 10.1093/ajcn/69.4.773S. PMID 10195602
- [Background] Weber JL, Cunningham-Sabo L, Skipper B, Lytle L, Stevens J, Gittelsohn J, Anliker J, Heller K, Pablo JL. Portion-size estimation training in second- and third-grade American Indian children. Am J Clin Nutr. 1999 Apr;69(4 Suppl):782S-787S. doi: 10.1093/ajcn/69.4.782S. PMID 10195603
- [Background] Going SB, Levin S, Harrell J, Stewart D, Kushi L, Cornell CE, Hunsberger S, Corbin C, Sallis J. Physical activity assessment in American Indian schoolchildren in the Pathways study. Am J Clin Nutr. 1999 Apr;69(4 Suppl):788S-795S. doi: 10.1093/ajcn/69.4.788S. PMID 10195604
- [Background] Davis SM, Going SB, Helitzer DL, Teufel NI, Snyder P, Gittelsohn J, Metcalfe L, Arviso V, Evans M, Smyth M, Brice R, Altaha J. Pathways: a culturally appropriate obesity-prevention program for American Indian schoolchildren. Am J Clin Nutr. 1999 Apr;69(4 Suppl):796S-802S. doi: 10.1093/ajcn/69.4.796S. PMID 10195605
- [Background] Snyder P, Anliker J, Cunningham-Sabo L, Dixon LB, Altaha J, Chamberlain A, Davis S, Evans M, Hurley J, Weber JL. The Pathways study: a model for lowering the fat in school meals. Am J Clin Nutr. 1999 Apr;69(4 Suppl):810S-815S. doi: 10.1093/ajcn/69.4.810S. PMID 10195607
- [Background] Helitzer DL, Davis SM, Gittelsohn J, Going SB, Murray DM, Snyder P, Steckler AB. Process evaluation in a multisite, primary obesity-prevention trial in American Indian schoolchildren. Am J Clin Nutr. 1999 Apr;69(4 Suppl):816S-824S. doi: 10.1093/ajcn/69.4.816S. PMID 10195608
- [Background] Stevens J, Story M, Becenti A, French SA, Gittelsohn J, Going SB, Juhaeri, Levin S, Murray DM. Weight-related attitudes and behaviors in fourth grade American Indian children. Obes Res. 1999 Jan;7(1):34-42. doi: 10.1002/j.1550-8528.1999.tb00388.x. PMID 10023728
- [Background] Gittelsohn J, Evans M, Helitzer D, Anliker J, Story M, Metcalfe L, Davis S, Iron Cloud P. Formative research in a school-based obesity prevention program for Native American school children (Pathways). Health Educ Res. 1998 Jun;13(2):251-65. doi: 10.1093/her/13.2.251. PMID 10181023
- [Background] Koehler KM, Cunningham-Sabo L, Lambert LC, McCalman R, Skipper BJ, Davis SM. Assessing food selection in a health promotion program: validation of a brief instrument for American Indian children in the southwest United States. J Am Diet Assoc. 2000 Feb;100(2):205-11. doi: 10.1016/S0002-8223(00)00064-X. PMID 10670393
- [Background] Teufel NI, Perry CL, Story M, Flint-Wagner HG, Levin S, Clay TE, Davis SM, Gittelsohn J, Altaha J, Pablo JL. Pathways family intervention for third-grade American Indian children. Am J Clin Nutr. 1999 Apr;69(4 Suppl):803S-809S. doi: 10.1093/ajcn/69.4.803S. PMID 10195606
- [Background] Davis SM, Reid R. Practicing participatory research in American Indian communities. Am J Clin Nutr. 1999 Apr;69(4 Suppl):755S-759S. doi: 10.1093/ajcn/69.4.755S. PMID 10195598
- [Background] Story M, Stevens J, Evans M, Cornell CE, Juhaeri, Gittelsohn J, Going SB, Clay TE, Murray DM. Weight loss attempts and attitudes toward body size, eating, and physical activity in American Indian children: relationship to weight status and gender. Obes Res. 2001 Jun;9(6):356-63. doi: 10.1038/oby.2001.46. PMID 11399782
- [Background] Lohman TG, Caballero B, Himes JH, Davis CE, Stewart D, Houtkooper L, Going SB, Hunsberger S, Weber JL, Reid R, Stephenson L. Estimation of body fat from anthropometry and bioelectrical impedance in Native American children. Int J Obes Relat Metab Disord. 2000 Aug;24(8):982-8. doi: 10.1038/sj.ijo.0801318. PMID 10951536
- [Background] Thompson JL, Davis SM, Gittelsohn J, Going S, Becenti A, Metcalfe L, Stone E, Harnack L, Ring K. Patterns of physical activity among American Indian children: an assessment of barriers and support. J Community Health. 2001 Dec;26(6):423-45. doi: 10.1023/a:1012507323784. PMID 11759094
- [Background] Hunsberger S, Murray D, Davis CE, Fabsitz RR. Imputation strategies for missing data in a school-based multi-centre study: the Pathways study. Stat Med. 2001 Jan 30;20(2):305-16. doi: 10.1002/1097-0258(20010130)20:23.0.co;2-m. PMID 11169604
- [Background] Story M, Snyder P, Anliker J, Cunningham-Sabo L, Weber JL, Platero H, Stone EJ. Nutrient content of school meals in elementary schools on American Indian reservations. J Am Diet Assoc. 2002 Feb;102(2):253-6. doi: 10.1016/s0002-8223(02)90060-x. No abstract available. PMID 11846122
- [Background] Lytle LA, Dixon LB, Cunningham-Sabo L, Evans M, Gittelsohn J, Hurley J, Snyder P, Stevens J, Weber J, Anliker J, Heller K, Story M. Dietary intakes of Native American children: findings from the pathways feasibility study. J Am Diet Assoc. 2002 Apr;102(4):555-8. doi: 10.1016/s0002-8223(02)90129-x. No abstract available. PMID 11985417
- [Background] Caballero B, Clay T, Davis SM, Ethelbah B, Rock BH, Lohman T, Norman J, Story M, Stone EJ, Stephenson L, Stevens J; Pathways Study Research Group. Pathways: a school-based, randomized controlled trial for the prevention of obesity in American Indian schoolchildren. Am J Clin Nutr. 2003 Nov;78(5):1030-8. doi: 10.1093/ajcn/78.5.1030. PMID 14594792
- [Background] Caballero B, Himes JH, Lohman T, Davis SM, Stevens J, Evans M, Going S, Pablo J; Pathways Study Research Group. Body composition and overweight prevalence in 1704 schoolchildren from 7 American Indian communities. Am J Clin Nutr. 2003 Aug;78(2):308-12. doi: 10.1093/ajcn/78.2.308. PMID 12885714
- [Background] Story M, Snyder MP, Anliker J, Weber JL, Cunningham-Sabo L, Stone EJ, Chamberlain A, Ethelbah B, Suchindran C, Ring K. Changes in the nutrient content of school lunches: results from the Pathways study. Prev Med. 2003 Dec;37(6 Pt 2):S35-45. doi: 10.1016/j.ypmed.2003.08.009. PMID 14636807
- [Background] Gittelsohn J, Davis SM, Steckler A, Ethelbah B, Clay T, Metcalfe L, Rock BH. Pathways: lessons learned and future directions for school-based interventions among American Indians. Prev Med. 2003 Dec;37(6 Pt 2):S107-12. doi: 10.1016/j.ypmed.2003.08.001. PMID 14636815
- [Background] Gittelsohn J, Merkle S, Story M, Stone EJ, Steckler A, Noel J, Davis S, Martin CJ, Ethelbah B. School climate and implementation of the Pathways study. Prev Med. 2003 Dec;37(6 Pt 2):S97-106. doi: 10.1016/j.ypmed.2003.08.010. PMID 14636814
- [Background] Lohman T, Thompson J, Going S, Himes JH, Caballero B, Norman J, Cano S, Ring K. Indices of changes in adiposity in American Indian children. Prev Med. 2003 Dec;37(6 Pt 2):S91-6. doi: 10.1016/j.ypmed.2003.08.004. PMID 14636813
- [Background] Steckler A, Ethelbah B, Martin CJ, Stewart D, Pardilla M, Gittelsohn J, Stone E, Fenn D, Smyth M, Vu M. Pathways process evaluation results: a school-based prevention trial to promote healthful diet and physical activity in American Indian third, fourth, and fifth grade students. Prev Med. 2003 Dec;37(6 Pt 2):S80-90. doi: 10.1016/j.ypmed.2003.08.002. PMID 14636812
- [Background] Stevens J, Story M, Ring K, Murray DM, Cornell CE, Juhaeri, Gittelsohn J. The impact of the Pathways intervention on psychosocial variables related to diet and physical activity in American Indian schoolchildren. Prev Med. 2003 Dec;37(6 Pt 2):S70-9. doi: 10.1016/j.ypmed.2003.08.012. PMID 14636811
- [Background] Going S, Thompson J, Cano S, Stewart D, Stone E, Harnack L, Hastings C, Norman J, Corbin C. The effects of the Pathways Obesity Prevention Program on physical activity in American Indian children. Prev Med. 2003 Dec;37(6 Pt 2):S62-9. doi: 10.1016/j.ypmed.2003.08.005. PMID 14636810
- [Background] Himes JH, Ring K, Gittelsohn J, Cunningham-Sabo L, Weber J, Thompson J, Harnack L, Suchindran C. Impact of the Pathways intervention on dietary intakes of American Indian schoolchildren. Prev Med. 2003 Dec;37(6 Pt 2):S55-61. doi: 10.1016/j.ypmed.2003.08.003. PMID 14636809
- [Background] Gunnarsson LG, Bodin L, Soderfeldt B, Axelson O. A case-control study of motor neurone disease: its relation to heritability, and occupational exposures, particularly to solvents. Br J Ind Med. 1992 Nov;49(11):791-8. doi: 10.1136/oem.49.11.791. PMID 1463680
- [Background] Stone EJ, Norman JE, Davis SM, Stewart D, Clay TE, Caballero B, Lohman TG, Murray DM. Design, implementation, and quality control in the Pathways American-Indian multicenter trial. Prev Med. 2003 Dec;37(6 Pt 2):S13-23. doi: 10.1016/j.ypmed.2003.08.006. PMID 14636805
- [Background] Story M, Stevens J, Himes J, Stone E, Rock BH, Ethelbah B, Davis S. Obesity in American-Indian children: prevalence, consequences, and prevention. Prev Med. 2003 Dec;37(6 Pt 2):S3-12. doi: 10.1016/j.ypmed.2003.08.008. PMID 14636804
- [Background] Cunningham-Sabo L, Snyder MP, Anliker J, Thompson J, Weber JL, Thomas O, Ring K, Stewart D, Platero H, Nielsen L. Impact of the Pathways food service intervention on breakfast served in American-Indian schools. Prev Med. 2003 Dec;37(6 Pt 2):S46-54. doi: 10.1016/j.ypmed.2003.08.007. PMID 14636808
- [Background] Weber JL, Lytle L, Gittelsohn J, Cunningham-Sabo L, Heller K, Anliker JA, Stevens J, Hurley J, Ring K. Validity of self-reported dietary intake at school meals by American Indian children: the Pathways Study. J Am Diet Assoc. 2004 May;104(5):746-52. doi: 10.1016/j.jada.2004.02.029. PMID 15127059